CLINICAL TRIAL: NCT03850977
Title: Association Between Chronic Pancreatitis and Respiratory Dysfunction: A Prospective Cohort Study?
Brief Title: Is There an Association Between Chronic Pancreatitis and Pulmonary Function
Acronym: RespPanc
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lise Gluud, Physician, PhD, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-18016860
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pancreatitis; Respiratory Insufficiency; Cirrhosis, Liver; Lung Function Decreased; Healthy
MeSH Terms: conditions — Pancreatitis, Chronic; Respiratory Insufficiency; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients and controls: Patients diagnosed with chronic pancreatitis or cirrhosis and healthy controls

SUMMARY:
To evaluate pulmonary function in chronic pancreatitis compared with healthy volunteers and patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pancreatitis or cirrhosis
* Healthy controls

Exclusion Criteria:

* Lack of informed consent
* Known chronic lung disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to include patients with chronic pancreatitis, cirrhosis and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Diffusion capacity of the lung for carbon monoxide | Three years
  Lung diffusion capacity
Alveolar volume | Three years
  Alveolar volume

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided